CLINICAL TRIAL: NCT02651870
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of a Combination Therapy of Candesartan and Amlodipine Versus Candesartan Monotherapy in Hypertensive Patients Inadequately Controlled by Candesartan Monotherapy
Brief Title: Trial to Evaluate the Efficacy and Safety of a Combination Therapy of Candesartan and Amlodipine Versus Candesartan Monotherapy in Hypertensive Patients Inadequately Controlled by Candesartan Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 144HT14020
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — candesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Candesartan 16mg + Amlodipine 5mg (Experimental): Candesartan 16mg + Amlodipine 5mg, po, q.d.
  Interventions: Drug: Candesartan 16mg; Drug: Amlodipine 5mg
- Candesartan 16mg + Amlodipine 10mg (Experimental): Candesartan 16mg + Amlodipine 10mg, po, q.d.
  Interventions: Drug: Candesartan 16mg; Drug: Amlodipine 10mg
- Candesartan 16mg (Active Comparator): Candesartan 16mg, po, q.d.
  Interventions: Drug: Candesartan 16mg

INTERVENTIONS:
Drug: Candesartan 16mg
Drug: Amlodipine 5mg
  Arms: Candesartan 16mg + Amlodipine 5mg
Drug: Amlodipine 10mg
  Arms: Candesartan 16mg + Amlodipine 10mg

SUMMARY:
A Phase 3 Trial to Evaluate the Efficacy and Safety of a Combination Therapy of Candesartan and Amlodipine Versus Candesartan Monotherapy in Hypertensive Patients Inadequately Controlled by Candesartan Monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 or above
* Inadequately controlled Essential hypertension at Screening

  1. Drug naive or didn't take antihypertensive drug within 2 weeks prior to Visit 1

     * Mean sitDBP ≥ 95mmHg on target arm
  2. Taking antihypertensive drug but not controlled

     * Mean sitDBP ≥ 90mmHg on target arm
* Inadequately controlled after 4 weeks of Candesartan 16mg monotherapy

  * Mean sitDBP at Visit 2 ≥ 90mmHg on target arm
* Ability to provide written informed consent

Exclusion Criteria:

* The change of mean sitDBP ≥ 10mmHg or mean sitSBP ≥ 20mmHg on target arm at Visit 1
* Mean sitDBP ≥ 120mmHg or mean sitSBP ≥ 200mmHg on target arm at Visit 1 and Visit 2
* Known to suspected Stage 2 Hypertension(aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* Patient with congestive heart failure(NYHA class III, IV)
* Patient with unstable angina pectoris, myocardial infarction, Valvular heart disease, arrhythmia(treatment required) within 3 months
* History of stroke, cerebral hemorrhage within 6 months
* Type I Diabetes mellitus, Type II Diabetes mellitus with HbA1c > 8.5%
* History of severe or malignant retinopathy
* AST/ALT > UNL*3, Serum creatinine > UNL*1.5, K > 5.5mEq/L
* Patient with acute or chronic inflammatory(treatment required) status
* Patient who need to take antihypertensive drug besides Investigational products
* Patient must be treated with medications prohibited for concomitant use during the study period
* History of angioedema related to ACE inhibitor or angiotensin II receptor blockers
* Hypersensitive to Candesartan/Amlodipine
* Patient who are dependent on drugs or alcohol within 6 months
* History of disability to drug ADME, active inflammatory bowel syndrome within 12months, impaired pancreatic function, GI bleeding, obstructions of urinary tract
* Patients treated with other investigational product within 30 days at first time taking the investigational product
* Women with pregnant, breast-feeding
* History of malignant tumor within 5 years
* Not eligible to participate for the study at the discretion of investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2016-02-25 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
The mean change of sitDBP(sitting diastolic blood pressure) | From baseline at week 8

SECONDARY OUTCOMES:
The mean change of sitDBP | From baseline to week 4
The mean change of sitSBP | From baseline to week 4 and 8
Control rate: Patient achieving sitSBP < 140mmHg and sitDBP < 90mmHg | From baseline to week 8
Response rate: sitSBP reduction ≥ 20mmHg and sitDBP reduction ≥ 10mmHg | From baseline to week 8

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea